CLINICAL TRIAL: NCT00975728
Title: High Total Antioxidant Capacity (TAC) Products Added to Diet: Clinical and Instrumental Evaluation of Their Effect on Skin Surface Parameters and on Photo-induced Acute Damage of the Skin (Double Blind Clinical Study vs Placebo)
Brief Title: High Total Antioxidant Capacity Products Added to Diet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Derming SRL (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Adele Sparavigna, DermIng S.r.l.
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DermIng E0709
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: Anti-oxidant; Açai; Food supplement; Sun protection; Skin erythema prevention; Anti-oxidant efficacy; Anti-age efficacy; Skin photo-induced damage protection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 Product 825 (2-servings day) (Experimental): 30 subjects drinking 2 servings day of Product 825 for 8 weeks
  Interventions: Dietary Supplement: Alixir - Pomegranate, apple and Açai drink / Placebo
- Group 1 Product 824 (2 servings-day) (Experimental): 30 subjects drinking 2 servings-day of Product 824 for 8 weeks
  Interventions: Dietary Supplement: Alixir - Pomegranate, apple and Açai drink / Placebo
- Group 2 Product 825 (1 serving-day) (Experimental): 30 subjects drinking 1 serving-day of Product 825 for 8 weeks
  Interventions: Dietary Supplement: Alixir - Pomegranate, apple and Açai drink / Placebo
- Gruop 2 Product 824 (1 serving-day) (Experimental): 30 subjects drinking 1 serving-day of Product 824 for 8 weeks
  Interventions: Dietary Supplement: Alixir - Pomegranate, apple and Açai drink / Placebo

INTERVENTIONS:
Dietary Supplement: Alixir - Pomegranate, apple and Açai drink / Placebo — 250 ml/day Alixir/Placebo for Group 2 for 8 weeks 500 ml/day Alixir/Placebo for Group 1 for 8 weeks
  Other Names: Barilla Alixir (code 824/825); Anti-oxidant drink; Açai drink

SUMMARY:
The purpose of this study is to evaluate the antioxidant activity on skin photo induced damage of a food supplement and its anti-age properties.

DETAILED DESCRIPTION:
To determine the antioxidant activity of the tested product the following clinical and instrumental evaluations will be performed:

1. Evaluation of experimentally induced erythema inhibition: in basal conditions, before starting the assumption of the test product/placebo, and at T4, T8, T12, T16 weeks, each volunteer wll be exposed at the level of dorsal skin to six incremental doses of UVR (ultraviolet radiations mJ/cm2 ) in order to determine the MED (minimal erythema dose of unprotected skin). 20+/-4 hours after the UV exposure clinical and instrumental (optical densitometry) evaluations of skin erythema and photographic documentation (only on 16 preselected cases) will be performed.
2. Blood samples collection for the determination of the principal antioxidants concentration (for example: lutein, carotene, lycopene and E vitamin): at T0, T4, T8 and T12 blood samples (5 ml of venous blood) will be collected on each volunteer by the Medical Staff. The samples will be sent to an external laboratory for haematologic control task.

To determine the anti-age properties of the tested product the following clinical and instrumental evaluations will be performed:

1. Non Invasive, instrumental evaluation of principal skin parameters: epicutaneous pH, skin hydration (skin electrical capacitance), skin firmness (plastoelasticity), skin texture (skin surface irregularity index - FFT on skin replicas) measurements will be performed at T0 and T8 mono-laterally at level of volar forearm medium third, left or right side according to a previously defined randomization list.
2. Clinical pictures with UV flash (Wood's light): at T0 and T8, 20 preselected cases of fairy skinned volunteers (selected on the basis of clinical ananmnesis regarding photosensitivity) will be submitted to the realization of clinical pictures at the level of the face using a special UV flash, able to highlight melanin spots, even if not yet visible at the naked eye.

Moreover aim of the study is also to evaluate the best dosage of the beverage (1 or 2 servings of 250 ml/a day).

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers of both sexes, between 30 and 60 years of age
* Phototype II or III ( Fitzpatrick's classification)
* Volunteers in a good general state of health in the Investigator opinion
* Volunteers not taking drugs or undergoing surgical procedure
* Volunteers who are giving a written informed consent

Exclusion Criteria:

* pregnancy
* lactation
* smoking >10 cigarettes per day
* drinking more then one glass of wine per day
* drinking super-alcoholics
* assumption of food supplement
* change in the normal habits in the last month
* participation in a similar study during the previous 3 months
* insufficient adhesion to the study protocol
* dermatological disease
* clinical and significant skin condition on the test area (e.g. lesions, scars,malformations)
* diabetes
* endocrine disease
* hepatic, renal or cardiac disorder
* cancer
* topical drugs or surgical procedure on the test areas during the previous 3 months
* systemic corticosteroids
* aspirin or non-steroid anti-inflammatory drugs (FANS)
* diuretic drugs
* antibiotics and chemotherapics
* psychotropic drugs
* retinoids
* psoralens
* cardiologic and vascular drugs

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Erythema evaluation (MED-optical densitometry) | T0 (basal conditions), T4 and T8 (after 4 and 8 week-treatment), T12 and T16 (follow-up visits - 12 and 16 weeks after T0)

SECONDARY OUTCOMES:
Skin evaluations (Skin texture - Hydration - Plastoelasticity - Epicutaneous pH) | T0 and T8 for skin evaluations - T0, T4, T8 and T12 for blood analysis
Determination on blood samples of antioxidants diet components | T0 and T8 for skin evaluations - T0, T4, T8 and T12 for blood analysis

CONTACTS AND LOCATIONS:
Overall Officials: Adele Sparavigna, Doctor, Principal Investigator — Derming SRL
Locations (1):
- DermIng S.r.l, Monza, MB, Italy

REFERENCES:
- [Background] Elsner P., Berardesca E., Maibach H. Bioengineering of the skin: Water and the stratum corneum CRC Press, Boca Raton, 1994; Fuga GC, Spina C, Cavallotti C, Di Palma A, Lombardi G, Marmo W Computerized reflected optical densitometry. A research on the colour of the skin - Journal of Applied Cosmetology, 8:91-110,1990; Cosmetic, Toiletry and Fragrance Association of South Africa (CFTA), The European Cosmetic Toiletry and Perfumery Association (COLIPA), Japan Cosmetic Industry Association (JCIA) International sun protection factor (SPF) test method; October 2002; ICH Harmonised Tripartite Guideline - Guideline for Good Clinical Practice International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use: May 1996; Setaro M., Sparavigna A. Morphological Evaluation of Skin Surface by Fourier's Transform: A Study on the Phase and the Modulus
- See also: Investigator center — http://www.derming.com
- See also: Sponsor — http://www.barilla.it
- See also: Haematological laboratory center — http://www.biochimica.unibo.it/Biochimica/default.htm